CLINICAL TRIAL: NCT07002281
Title: A Single-center, Open-label, Single-dose Clinical Trial to Evaluate the Absorption, Metabolism, and Excretion of 3 mg/100 μCi [14C]Azvudine Suspension in Vivo in Healthy Male Subjects
Brief Title: [14C] Mass Balance Clinical Trial of Azvudine in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GQ-FNC-111
Record Dates: First submitted 2025-05-13; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Azvudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy male subjects (Experimental)
  Interventions: Drug: [14C]Azvudine suspension

INTERVENTIONS:
Drug: [14C]Azvudine suspension — A single oral dose of 3 mg/100 μCi of [14C]Azvudine suspension is given orally on an empty stomach.

SUMMARY:
Azvudine(FNC)，a nucleoside reverse transcriptase inhibitor, make itself a better candidate to be co-formulated in other anti-HIV therapies, thus to improve patient's compliance. FNC is a broad-spectrum RNA virus inhibitor that inhibits the novel coronavirus RNA-dependent RNA polymerase (RdRp).

This trial uses a single-center, open-label, single-dose adaptive design aimed at investigating the pharmacokinetic characteristics of total radioactivity of [14C]-labeled Azvudine in whole blood and plasma of healthy male subjects, to quantitatively analyze the total radioactivity in exhaled gas and excreta of healthy male subjects after oral administration of [14C]Azvudine suspension, to obtain data on the mass balance in the human body, and to determine the main excretion routes. Biological sample collection and safety examination will be performed in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male subjects aged 18~45 years old;
2. Body mass index (BMI) within the range of 18.0-30.0 (including the critical value) (BMI = weight (kg) / height 2 (m2)), the weight should be ≥ 50.0kg;
3. Subjects who are judged by the investigator to be in good health, with normal results of physical examination, vital signs, electrocardiogram, and laboratory examinations or abnormal but without clinical significance;
4. Subjects who have no fertility plan during the study period and within 1 year after the end of the trial and agree to take effective non-drug contraceptive measures during the trial (except for those who have taken permanent contraceptive measures, such as vasectomy, etc.), and have no sperm donation plan;
5. Subjects who are willing to follow the visits, study treatments, laboratory tests, and other study-related procedures and requirements specified in the study protocol, understand and sign the informed consent form.

Exclusion Criteria:

1. Those who are allergies, with a history of drug or food allergies, especially those who are allergic to any of the ingredients in this product and excipients;
2. Those who are positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab), or treponema pallidum antibody;
3. Those who cannot tolerate venipuncture blood collection and/or have a history of blood sickness and needle sickness;
4. Those who have a history of mental illness, family history of mental illness, or chronic or serious diseases of the central nervous system, cardiovascular, liver, kidney, lung, metabolic, blood, bone and other systems;
5. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5 times the upper limit of normal (ULN);
6. Glomerular filtration rate< 90 mL/min/1.73m2;
7. Patients with long QT syndrome or its family history, or QTcF interval (Fridericia's correction) > 450 ms; Intraventricular block or left and right bundle branch block and/or QRS>120 ms; Frequent ventricular ectopic beats (1 premature ventricular contraction occurred on any 10-second ECG during the screening period≥); or abnormal resting heart rate (>100 bpm);
8. Previous or current swallowing dysfunction, active gastrointestinal diseases (such as chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease) or other diseases that significantly affect drug absorption, distribution, metabolism and excretion;
9. Hemorrhoids or perianal disease accompanied by regular/hematochezia;
10. Those who have donated blood within 3 months before screening, or have lost ≥ 200 ml of blood, or plan to donate blood during the study period;
11. Those who have been vaccinated with the new crown vaccine within 2 weeks before screening or other vaccines within 3 months before screening or plan to be vaccinated during the trial;
12. Intake of > 6 servings of coffee, tea, cola, energy drinks, or other caffeinated products per day within 3 months prior to screening (one serving ≈ 120 mg of caffeine); or ingestion of foods or drinks containing high levels of caffeine, xanthines, alcohol, flavonoids (such as: grapefruit (juice), grapefruit (juice), orange (juice), etc.) within 24 hours before administration;
13. Use of any drug that inhibits or induces hepatic drug metabolism enzymes within 1 month before administration (such as: inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; Inhibitors - SSRIs antidepressants, cimetidine, diltiazem macrolides, nitroimidazoles, sedative-hypnotics, verapamil, fluoroquinolones, antihistamines, etc.);
14. Have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, and health care products within 14 days before administration;
15. Those who have participated in other clinical trials within 3 months before screening;
16. Smoking more than 5 cigarettes per day within 3 months before screening, or unable to comply with the prohibition of smoking during the study;
17. Those who have a history of alcoholism within 12 months before screening (drinking ≥ 14 units of alcohol per week: 1 unit = 360 mL of beer, or 45 mL of spirits, or 150 mL of wine) or those who have a positive alcohol breath test before enrollment;
18. Known or suspected history of drug abuse (e.g., morphine, methamphetamine, ketamine, methylenedioxyamphetamine, tetrahydrocannabinolic acid, cocaine, etc.), or positive test for addictive substances;
19. Surgical surgery within 3 months prior to screening, or planned surgical surgery during the current study period;
20. Participated in radiolabeled clinical trials within 1 year before screening;
21. Workers who require long-term exposure to radioactive conditions, or who have had significant radioactive exposure within 1 year before the test (≥ 2 chest/abdominal CT examinations, or ≥ 3 other types of X-ray examinations);
22. The investigator judges that there are other circumstances that make subjects unsuitable to participate in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of total radioactive material in whole blood and plasma | Up to 96 hours post-dose
Pharmacokinetics (PK): Time to Maximum Concentration (Tmax) of total radioactive material in whole blood and plasma | Up to 96 hours post-dose
Pharmacokinetics (PK): Area Under the Concentration curve (AUC) of total radioactive material in whole blood and plasma | Up to 96 hours post-dose
Pharmacokinetics (PK): Elimination half-life (t1/2) of total radioactive material in whole blood and plasma | Up to 96 hours post-dose
The total radioactivity allocation ratio | Up to 96 hours post-dose
The total radioactivity and the percentage to the total administered dose | Up to 168 hours post-dose

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of Azvudine and its metabolites in plasma | Up to 96 hours post-dose
Pharmacokinetics (PK): Time to Maximum Concentration (Tmax) of Azvudine and its metabolites in plasma | Up to 96 hours post-dose
Pharmacokinetics (PK): Area Under the Concentration curve (AUC) of Azvudine and its metabolites in plasma | Up to 96 hours post-dose
Pharmacokinetics (PK): Elimination half-life (t1/2) of Azvudine and its metabolites in plasma | Up to 96 hours post-dose
Percentage of Azvudine metabolites in plasma to total exposed AUC | Up to 96 hours post-dose
Occurrence of Adverse Events | From enrollment to the end of the study on Day 22.
  Clinical presentation characteristics, severity, onset time, duration of adverse events, management measures, outcomes, and the correlation with the investigational drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan Hospital, Beijing, China